CLINICAL TRIAL: NCT04462965
Title: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of Toripalimab Combined With Temozolomide and Cisplatin in the Postoperative Adjuvant Treatment of Completely Resected Mucosal Melanoma
Brief Title: Postoperative Adjuvant Treatment of Completely Resected Mucosal Melanoma Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Associate Director of Beijing University Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-ISS-CO148
Record Dates: First submitted 2020-05-28; First posted 2020-07-08 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Mucosal Melanoma
MeSH Terms: interventions — toripalimab; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Toripalima Combined with Temozolomide and Cisplatin. Toripalima3 mg/kg intravenous infusion, administered once every 2 weeks (1 treatment cycle every 2 weeks) for a maximum of 1 year. Temozolomide, Oral 200mg/m2 1-5 days and Cisplatin, Iv infusion 25 mg/m2/d for a period of 1 to 3 days, 28 days for 1 cycle, lasting 6 cycles;
  Interventions: Combination Product: Toripalimab
- Placebo group (Placebo Comparator): Placebo Combined with Temozolomide and Cisplatin. Toripalima3 mg/kg intravenous infusion, administered once every 2 weeks (1 treatment cycle every 2 weeks) for a maximum of 1 year. Temozolomide, Oral 200mg/m2 1-5 days and Cisplatin, Iv infusion 25 mg/m2/d for a period of 1 to 3 days, 28 days for 1 cycle, lasting 6 cycles;
  Interventions: Combination Product: Temozolomide

INTERVENTIONS:
Combination Product: Toripalimab — Injection,Specification 240mg/6ml, 3 mg/kg for the dose, iV, every 2 weeks a dose cycle, up to 1 year; Temozolomide: 100mg or 20mg, Every 4 weeks a dose cycle, up to 6 cycles Cisplatin: Injection, 20mg,Every 4 weeks a dose cycle, up to 6 cycles
  Arms: Test group
Combination Product: Temozolomide — Placebo：Injection,Specification 240mg/6ml, 3 mg/kg for the dose, iV, every 2 weeks a dose cycle, up to 1 year; Temozolomide: 100mg or 20mg, Every 4 weeks a dose cycle, up to 6 cycles Cisplatin: Injection, 20mg,Every 4 weeks a dose cycle, up to 6 cycles
  Arms: Placebo group

SUMMARY:
A mucosal melanoma postoperative adjuvant treatment of multicenter, randomized, double-blind, placebo-controlled phase II study, evaluation of mucosal melanoma patients accept completely resected, Toripalima Combined with Temozolomide and Cisplatin postoperative adjuvant therapy efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female；
2. Histopathologically confirmed and diagnosed as mucosal melanoma;
3. ECOG score 0 or 1;
4. The primary lesion is completely resected and the surgical margin is (-); Complete whole-body staging examination (including: brain enhanced CT or MRI, chest, abdomen, pelvic enhanced CT (nasopharyngeal MRI or CT, oropharyngeal MRI or CT), superficial lymph node b-ultrasound; or whole body PET-CT) should be performed before enrollment to confirm there are no regional or distant metastases (patients with contrast media allergy may choose plain CT);
5. The patient is not receiving standard adjuvant treatment；
6. No contraindications, having adequate organ and marrow function；
7. Use of highly-effective contraceptive methods during the whole study for men of reproduction ability or women of childbearing potential (e.g. oral contraceptives, intrauterine contraceptive device, abstinence of sexual intercourse or barrier contraception in combination with spermatocide), and continuation of contraception for 12 months after the end of treatment；
8. Enrolled for treatment within 4 months post-procedure;
9. The subject is voluntary to participate in the study, sign the informed consent form, with good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2;
2. Known allergy to recombinant humanized anti-PD-1 monoclonal antibody drug and its components;
3. High dose of interferon therapy or adjuvant chemotherapy (Temozolomide + Cisplatin) was performed after surgery;
4. Skin melanoma, eye melanoma(except the conjunctival), melanoma with unknown primary foci;
5. The primary lesion is not completely resected;
6. Staging examination indicated residual or metastatic tumor;
7. Female patients who are pregnant or lactating, or of childbearing potential but not using appropriate contraceptive measures;
8. Currently having serious and uncontrolled acute infection; or suppurative infection and chronic infection with prolonged wound healing;
9. Having serious heart disorder, including cardiac failure congestive, uncontrollable high-risk arrhythmia, unstable angina pectoris, infarct myocardial, severe cardiac valve disease and refractory hypertension;
10. Having neurological, mental disease or mental disorder that can not be easily controlled, poor compliance, inability to cooperate and narrate therapeutic response;
11. Patients with other malignant tumors at the same time;
12. Patients paticipated in other clinical trials at the same time;
13. Positive HIV; positive HCV; positive HBsAg or HBcAb whilst positive HBV DNA copies detected (limit of quantitation 500 IU/mL);
14. Active autoimmune diseases requiring systemic treatment in the past two years (e.g., use of disease-regulating drug, corticosteroid or immunosuppressant), relevant replacement therapy is allowed (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for renal or pituitary insufficiency);
15. Having received live vaccine within 4 weeks prior to the start of treatment;
16. Other severe, acute or chronic medical diseases or mental diseases or abnormalities in laboratory examination possibly increasing the relevant risk in study participation or possibly interfering the interpretation of study results as judged by the investigators..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
RFS assessment per RECIST 1.1. | 2 years
  To Compare the recurrence free survival (RFS) per response evaluation crieria in solid tumors(RECIST 1.1) in subjects of the postoperative adjuvant treatment of completely resected mucosal melanoma treated between Toripalima combined with Temozolomide and Cisplatin and placebo combined with Temozolomideand Cisplatin .

SECONDARY OUTCOMES:
RFS assessment per RECIST1.1 in 1 year and 2 year; | 2 years
  1 year and 2 year recurrence free survival rate of completely resected mucosal melanoma with postoperative adjuvant treatment, will be assessed using RECIST1.1 to evaluate tumor recurrence.
DMFS assessed by investigator per RECIT1.1; | 2 years
  Distant metastasis free survival (DMFS) of completely resected mucosal melanoma with postoperative adjuvant treatment per RECIST 1.1;
Overall survival (OS) per death time; | 2 years
  Overall survival (OS) of completely resected mucosal melanoma with postoperative adjuvant treatment per death time;
.Incidence and grade of AEs and SAEs related to study drugs per NCI-CTCAE version 5.0, AEs ≥ grade 3 related to the study drugs. | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 for safty evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China